CLINICAL TRIAL: NCT05378984
Title: Cocoa Intake and Muscle Pain Sensation: an Experimental Study
Brief Title: Cocoa Intake and Muscle Pain Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Nikolaos Christidis, Associate professor, senior lecturer, senior consultant, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CHIMPS
Record Dates: First submitted 2022-05-10; First posted 2022-05-18 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Muscle Pain
Keywords: Myalgia; Experimental pain; Human; Temporomandibular disorders; Cocoa
MeSH Terms: conditions — Myalgia; Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The chocolate given to the participant was of a different concentration of cocoa, distributed in a randomized and double-blinded order. The participants where given the chocolate with their eyes closed. A non-blinded examiner fed the chocolate to the participant at each clinical trial, while a blinded examiner did the assessments. The different types of chocolates were given at three different visits to all participants with at least one week of washout in between. To randomize the order in which the chocolates were given to each participant, an internet-based site was used (www.randomization.com; Seed 19525). The randomization was done in five blocks of six participants each, by a researcher who did not participate in the data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dark Chocolate (Active Comparator)
  Interventions: Other: before - hypertonic saline 5%; Other: after - hypertonic saline 5%
- Milk Chocolate (Active Comparator)
  Interventions: Other: before - hypertonic saline 5%; Other: after - hypertonic saline 5%
- White Chocolate (Active Comparator)
  Interventions: Other: before - hypertonic saline 5%; Other: after - hypertonic saline 5%

INTERVENTIONS:
Other: before - hypertonic saline 5% — pain was induced by intramuscular injections of hypertonic saline (5%)
Other: after - hypertonic saline 5% — pain was induced by intramuscular injections of hypertonic saline (5%)

SUMMARY:
This experimental randomized, double-blind, and controlled study included fifteen young, healthy, and pain-free men and 15 age-matched women.

It lasted for three visits with at least one-week washout. Pain was experimentally induced, twice at each visit, with intramuscular injections of 0.2 mL hypertonic saline (5%), before and after intake of one of the different chocolate-types; white (30% cocoa-content), milk (34% cocoa-content), dark (70% cocoa-content). Pain duration, pain area, peak pain, and pressure pain threshold were assessed every fifth minute after each injection, between the time-points 5 to 30 min.

Prior to inclusion, all participants underwent an examination in a dental chair. This included a clinical examination of the orofacial region according to the Diagnostic Criteria for temporomandibular disorders (DC/TMD) by a blinded examiner. Participants were also examined regarding their psychosocial status prior to inclusion, this included depression, somatization, anxiety, pain catastrophizing and stress.

ELIGIBILITY:
Inclusion Criteria:

1. good general health
2. age between 18-40 years

Exclusion Criteria:

1. any pain-related diagnosis of TMD or of the orofacial region
2. any headaches
3. a diagnosis of systemic muscular or joint diseases (fibromyalgia or rheumatoid arthritis)
4. whiplash-associated disorders
5. neurological disorders
6. psychiatric disorders
7. any allergy to the substances used

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity by intake of chocolate | 5 min after injection of hypertonic saline
  Pain intensity will be assssed using a 0-100 visual analoge scale (0-no pain; 100-worst pain ever experienced)
Change in peak pain intensity before and after intake of chocolate | 5 min after injection of hypertonic saline
  Peak pain intensity will be asessed from the 0-100 visual analoge scale (0-no pain; 100-worst pain ever experienced)
Change in pain duration by intake of chocolate | Pain duration up to 300 seconds after injection of hypertonic saline
  Pain duration is assessed in seconds.
Change in pain area by intake of chocolate | Pain area is marked 5 min after injection of hypertonic saline
  Pain area will be marked on lateral charts of the head before and after intake of chocolate and measured in au.

SECONDARY OUTCOMES:
Change in pressure pain threshold by intake of chocolate | Pressure pain thresholds are assessed 5 min after injection of hypertonic saline
  Pressure pain thresholds are assessed using a digital algometer over the area of injection in the masseter muscle with a pressure rate of 30kPa/s.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Department of Dental Medicine, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers upon request from any of the authors
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication and up to 20 years after publication
Access Criteria: Data will be shared with other researchers upon request from any of the authors

REFERENCES:
- [Derived] Hajati A, Brondani M, Angerstig L, Klein V, Liljeblad L, Al-Moraissi EA, Louca Jounger S, Brondani B, Christidis N. Chocolate intake and muscle pain sensation: A randomized experimental study. PLoS One. 2023 May 24;18(5):e0284769. doi: 10.1371/journal.pone.0284769. eCollection 2023. PMID 37224109